CLINICAL TRIAL: NCT06396260
Title: Structural and Functional Networks in ALS: An Insight Into Pseudobulbar Affect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Christian Holm Steenkjær, Principal Investigator, Aalborg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F2024-014
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Pseudobulbar Affect
Keywords: Diffusion Kurtosis Imaging; Magnetoencephalography; Connectivity
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Longitudinal imaging study. Baseline acquisition of DKI and resting state MEG of ALS and matched healthy controls. Participants with ALS will be monitored for a period of 6 months for symptoms of PBA. If developed, or not developed after 6 months, follow-up DKI and MEG will be acquired.
  An additional sub-study will be performed in patients with ALS and newly developed PBA, where resting state MEG will be acquired after at least 7 days of symptomatic treatment independent of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Sex- and age matched, healthy control. Will only have baseline DKI and MEG performed.
  Interventions: Other: Diffusion Kurtosis Imaging (DKI); Other: Resting State Magnetoencephalography
- ALS without PBA (Active Comparator): ALS patient without PBA, either at baseline and 6 month follow-up
  Interventions: Other: Diffusion Kurtosis Imaging (DKI); Other: Resting State Magnetoencephalography
- ALS with PBA (Active Comparator): ALS patient with PBA, either at baseline or follow-up
  Interventions: Other: Diffusion Kurtosis Imaging (DKI); Other: Resting State Magnetoencephalography

INTERVENTIONS:
Other: Diffusion Kurtosis Imaging (DKI) — Non-invasive MRI sequence which extracts information of diffusion signals from complex brain tissue
Other: Resting State Magnetoencephalography — Non-invasive method of measuring resting state brain activity through magnetoencephalography (MEG)

SUMMARY:
The investigators aim to elucidate characteristics of structural and functional brain connectivity in patients with amyotrophic lateral sclerosis (ALS) and pseudobulbar affect (PBA) using diffusion kurtosis imaging (DKI) and magnetoencephalography (MEG).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALS in the last 6 months according to Gold Coast Criteria

Exclusion Criteria:

* - Lack of ability to answer survey through own ability or through a surrogate, for example by hand controlled, eye-controlled computer and/or tablet, or through telephone interview.
* Lack of ability to cooperate.
* Pregnancy
* Drug addiction defined as the non-prescribed use of cannabis, opioids, or other narcotics.
* Alcohol addiction defined as over 21 units weekly.
* Lesional neurological diseases, such as stroke, tumor or multiple sclerosis
* Epilepsy
* Neurodegenerative diseases other than ALS
* Severe psychiatric disease such as major depression disorder, bipolar disease or schizophrenia
* Contraindication for MRI and MEG scan according to hospital guidelines
* Severe liver or kidney disease
* Dysregulated heart disease
* Ongoing treatment with any antidepressants or any antipsychotics at recruitment.
* Diagnosed with frontotemporal dementia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean kurtosis | Baseline measurement and up to 6 month follow-up measurements
  A measurement of kurtosis diffusion signal in pseudobulbar affect-affiliated brains areas (prefrontal lobe, pons, cerebellum, motor cortex, temporal lobe) derived from Diffusion kurtosis imaging (DKI)-MRI
Spectral connectivity | Baseline measurement and up to 6 month follow-up measurements
  Estimation of connectivity (correlation between spikes of activity) between pseudobulbar affect afflilated cortical brain areas (prefrontal cortex, motor cortex, temporal lobe) derived through resting state magnetoencelphalography (MEG)

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University hospital, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not planned to be available to other researchers. However findings from this study is planned to be published in peer-reviewed journal regardless of positive/negative findings